CLINICAL TRIAL: NCT00189449
Title: Effects of Long-Term Treatment With Nasally Inhaled Triamcinolone Acetonide in Children With Allergic Rhinitis
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Other Study IDs: IST Nasacort AQ NAS.US1.631; RC - 3421
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Allergic Rhinitis; Allergy; Growth
Keywords: Allergic Rhinitis; Allergy; Growth
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity

SUMMARY:
Seasonal/perennial allergic rhinitis (SAR/PAR) is a common childhood illness. One of the leading therapies for the treatment of SAR/PAR is intranasally inhaled corticosteroids (ICS). One of the major long-term safety concerns is whether ICS interferes with normal growth in allergic rhinitis children. Recent evidence suggests that nasal ICS may cause decreased growth. However, the effect of nasal ICS on long-term growth and the attainment of final adult height is unknown. Another potential systemic adverse effect of ICS use is suppression of the hypothalamic-pituitary-adrenal axis function. The primary hypothesis of this study is that triamcinolone acetonide aqueous nasal spray (TAA) will have no effect on measured adult height in relation to target adult height in children with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female aged 6-13 years of age
* Diagnosis of SAR/PAR, with symptoms within the past 3 months
* Positive skin test to inhalant allergen with negative saline control
* No previous use of intranasal inhaled, oral, IV or topical steroid use within past 6 months.
* If the subject has asthma, only mild intermittent (per NAPP) guidelines treated with PRN bronchodilator

Exclusion Criteria:

* screening height outside the 5th and 95th percentiles
* History of abnormal growth
* Any other chronic condition beside allergic rhinitis or mild intermittent asthma
* Subject who has insufficient allergic rhinitis symptoms to require daily therapy during the trial.
* Subject with a known hypersensitivity to any active ingredients or excipents in the study medications
* Subject with nasal candidiasis, acute or chronic sinusitis, significant nasal polyposis (impairs nasal breathing), or other gross anatomical deformity of the nose sufficient to impair nasal breathing (e.g., deviated septum)
* Subjects with a history of substance abuse, mental illness or retardation
* Subjects with a history or presence of glaucoma or posterior subcapsular cataract
* Subjects with nocturnal enuresis.
* Use of Theophylline, Intal/Tilade or leukotriene modifiers.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Study Completion 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: David Skoner, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States